CLINICAL TRIAL: NCT03019406
Title: An Open-label Ascending Dose Cohort Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of Avalglucosidase Alfa (NeoGAA, GZ402666) in Patients With Infantile-onset Pompe Disease Treated With Alglucosidase Alfa Who Demonstrate Clinical Decline or Sub-optimal Clinical Response
Brief Title: A Study to Assess Safety and Efficacy of Avalglucosidase Alfa Administered Every Other Week in Pediatric Patients With Infantile-onset Pompe Disease Previously Treated With Alglucosidase Alfa
Acronym: Mini-COMET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT14132; U1111-1179-4616 (Registry Identifier: ICTRP); 2016-003475-21 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2017-01-12 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Glycogen Storage Disease Type II-Pompe's Disease
MeSH Terms: interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Avalglucosidase Alfa 20 mg/kg (Experimental): Avalglucosidase alfa, 20 mg/kg intravenous (IV) infusion every other week (qow) for 25 weeks in the Primary Analysis Period (PAP), followed by same treatment from Week 26 up to Week 371 in extension treatment period (ETP).
  Interventions: Drug: Avalglucosidase alfa (GZ402666)
- Cohort 2: Avalglucosidase Alfa 40 mg/kg (Experimental): Avalglucosidase alfa 40 mg/kg IV infusion qow for 25 weeks in the PAP, followed by same treatment from Week 26 up to Week 371 in ETP.
  Interventions: Drug: Avalglucosidase alfa (GZ402666)
- Cohort 3a: Avalglucosidase Alfa 40 mg//kg (Experimental): After determination of the highest tolerated avalglucosidase alfa dose in Cohort 1 and Cohort 2 (after at least 5 participants in each Cohort 1 and Cohort 2 had received the 7th dose of avalglucosidase alfa or completed Week 13 with a minimum of 6 infusions), participants received avalglucosidase alfa 40 mg/kg (the highest tolerated dose) IV infusion qow for 25 weeks in PAP, followed by same treatment from Week 26 up to Week 371 in ETP.
  Interventions: Drug: Avalglucosidase alfa (GZ402666)
- Cohort 3b: Alglucosidase Alfa in PAP (Experimental): After determination of the highest tolerated avalglucosidase alfa dose in Cohort 1 and Cohort 2 (after at least 5 participants in each Cohort 1 and Cohort 2 had received the 7th dose of avalglucosidase alfa or completed Week 13 with a minimum of 6 infusions), participants received alglucosidase alfa at their current stable dose (defined as dose [between 20 mg/kg qow and 40 mg/kg weekly as per physician] administered regularly for a minimum of 6 months immediately prior to entry in this study) IV infusion for 25 weeks in PAP. After PAP, participants received avalglucosidase alfa 40mg/kg IV infusion qow from Week 26 up to Week 371 in ETP.
  Interventions: Drug: Avalglucosidase alfa (GZ402666); Drug: Alglucosidase alfa (GZ419829)

INTERVENTIONS:
Drug: Avalglucosidase alfa (GZ402666) — Pharmaceutical form: powder for concentrate for solution for infusion,
  Route of administration: IV
  Other Names: Nexviazyme
Drug: Alglucosidase alfa (GZ419829) — Pharmaceutical form: powder for concentrate for solution for infusion,
  Route of administration: IV
  Other Names: Myozyme®; Lumizyme®
  Arms: Cohort 3b: Alglucosidase Alfa in PAP

SUMMARY:
This is a multi-stage, phase 2, open-label, multicenter, multinational, ascending dose cohort, repeated intravenous (IV) infusion study of avalglucosidase alfa in pediatric patients with Infantile-Onset Pompe Disease (IOPD) who have been previously treated with alglucosidase alfa for a minimum of 6 months immediately prior to study entry and have demonstrated clinical decline or unsatisfactory clinical response.

DETAILED DESCRIPTION:
The duration of the study for each participant will be up to 9 years and 4 months that will consist of a 14-day screening period, that may be extended to up to 4 weeks in pre-specified situations. This is followed by a 25-week treatment period and an up to a 462-week treatment extension period and a 4-week post-treatment observation period. Cohort 1 and 2 (Cohort 1: avalglucosidase alfa 20 milligrams per kilogram [mg/kg], Cohort 2: avalglucosidase alfa 40 mg/kg) will be non-randomized and Cohort 3 (Cohort 3a: avalglucosidase alfa 40 mg/kg [maximum tolerated dose] and Cohort 3b: alglucosidase alfa) will be randomized.

ELIGIBILITY:
Inclusion criteria:

* The participants has confirmed acid alpha-glucosidase (GAA) enzyme deficiency from any tissue source.
* The participants who has reached legal age of majority as defined by local regulation, or the participant's legal guardian(s) must provide signed informed consent prior to performing any study-related procedures. If the participant is legally minor per local regulations, assent shall be obtained from participants, if applicable.
* The participants (and participant's legal guardian if participant is legally minor as defined by local regulation) must have the ability to comply with the clinical protocol.
* The participants is less than 18 years old.
* The participants, if female and of childbearing potential, must have a negative serum pregnancy test (beta-human chorionic gonadotropin) and must not breastfeeding at screening/Baseline.
* The participant has cardiomyopathy at the time of diagnosis: i.e., left ventricular mass index (LVMI) equivalent to mean age specific LVMI plus 2 standard deviations.
* The participant has been receiving a stable dose of alglucosidase alfa regularly for a minimum of 6 months immediately prior to study entry.
* For participants in Stage 1: The participant has documented evidence of clinical decline in at least 1 of the following parameters related to Pompe Disease and not related to intercurrent illness as assessed by the Investigator: respiratory function, motor skills, and/or cardiac parameters.
* For participants in Stage 2: The participant has documented evidence of suboptimal clinical response in at least 1 of the following parameters related to Pompe Disease and not related to intercurrent illness as assessed by the Investigator: respiratory function, motor skills, and/or new onset of ptosis.

Exclusion criteria:

Participants are excluded from the study if any of the following criteria apply:

* The participant has high antibody titer to alglucosidase alfa.
* The participant has a high risk for a severe allergic reaction to neoGAA (avalglucosidase alfa).
* The participant requires any prohibited concomitant medications (e.g., immune modulatory treatment) for the duration of the study.
* The participant has previously participated in any ACT14132 study cohort.
* Female participant of childbearing potential not protected by highly effective contraceptive method of birth control and/or who is unwilling or unable to tested for pregnancy.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2027-08-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- United States (3):
  - Regional Medical Genetics Center of New York Site Number : 8400002, Valhalla, New York
  - Duke University Medical Center Site Number : 8400001, Durham, North Carolina
  - Seattle Childrens Hospital and Regional Medical Center- Site Number : 8400005, Seattle, Washington
- France (4):
  - Investigational Site Number : 2500004, Nantes
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500002, Paris
  - Investigational Site Number : 2500001, Tours
- Japan (2):
  - Investigational Site Number : 3920001, Fuchu-shi, Tokyo
  - Investigational Site Number : 3920002, Fuchu-shi, Tokyo
- Investigational Site Number : 1580001, Hsinchu, Taiwan
- United Kingdom (2):
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260002, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kronn D, Davison J, Broomfield A, Brassier A, Labarthe F, Hahn SH, Kumada S, Ohki H, Prakalapakorn SG, Wilson C, Haack KA, Huynh-Ba O, Richards S, Sparks S, Tammireddy S, Zhou T, Chien YH, Kishnani PS; Mini-COMET investigators. The Mini-COMET Clinical Trial: Safety and Efficacy of Avalglucosidase Alfa after 97 Weeks of Treatment in Children with Infantile-Onset Pompe Disease Previously Treated with Alglucosidase Alfa. J Pediatr. 2025 Oct;285:114664. doi: 10.1016/j.jpeds.2025.114664. Epub 2025 May 29. PMID 40449831
- [Derived] Kishnani PS, Kronn D, Brassier A, Broomfield A, Davison J, Hahn SH, Kumada S, Labarthe F, Ohki H, Pichard S, Prakalapakorn SG, Haack KA, Kittner B, Meng X, Sparks S, Wilson C, Zaher A, Chien YH; Mini-COMET Investigators. Safety and efficacy of avalglucosidase alfa in individuals with infantile-onset Pompe disease enrolled in the phase 2, open-label Mini-COMET study: The 6-month primary analysis report. Genet Med. 2023 Feb;25(2):100328. doi: 10.1016/j.gim.2022.10.010. Epub 2022 Dec 21. PMID 36542086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 active centers in 5 countries. Total of 22 participants were screened between 12 October 2017 and 03 April 2019. None of the participants were screen failed. Participants were assigned to treatment by using interactive response technology system.
Pre-assignment Details: Participants in Cohorts 1 received avalglucosidase alfa 20 milligrams per kilogram (mg/kg) every other week (qow) and participants in Cohort 2 received avalglucosidase alfa 40 mg/kg qow. No randomization process was applied for Cohort 1 and 2. Participants in Cohort 3 were randomized (stratified by gender) to receive either avalglucosidase alfa 40 mg/kg qow (3a) or their current stable alglucosidase alfa dose regimen (3b). Data reported based on primary completion date, i.e., 30 September 2019.
Groups:
- Cohort 1: Avalglucosidase Alfa 20 mg/kg: Avalglucosidase alfa, 20 mg/kg intravenous (IV) infusion qow for 25 weeks in the Primary Analysis Period (PAP), followed by same treatment from Week 26 up to Week 371 in extension treatment period (ETP).
Period: PAP: up to 25 Weeks
Arm/Group | Cohort 1: Avalglucosidase Alfa 20 mg/kg | Cohort 2: Avalglucosidase Alfa 40 mg/kg | Cohort 3a: Avalglucosidase Alfa 40 mg//kg | Cohort 3b: Alglucosidase Alfa in PAP
Started | 6 | 5 | 5 | 6
Treated | 6 | 5 | 5 | 6
Completed | 6 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0
Period: ETP: Ongoing From Week 26
Arm/Group | Cohort 1: Avalglucosidase Alfa 20 mg/kg | Cohort 2: Avalglucosidase Alfa 40 mg/kg | Cohort 3a: Avalglucosidase Alfa 40 mg//kg | Cohort 3b: Alglucosidase Alfa in PAP
Started | 6 | 5 | 5 | 3 (Participants who completed PAP and accepted to receive avalglucosidase alfa treatment in ETP.)
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 5 | 5 | 3
Not completed — Ongoing | 6 | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included participants who had received at least 1 infusion (partial or total) and were analyzed according to treatment received.
Groups:
- Cohort 1: Avalglucosidase Alfa 20 mg/kg: Avalglucosidase alfa, 20 mg/kg IV infusion qow for 25 weeks in the PAP, followed by same treatment from Week 26 up to Week 371 in extension treatment period (ETP).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Avalglucosidase Alfa 20 mg/kg | Cohort 2: Avalglucosidase Alfa 40 mg/kg | Cohort 3a: Avalglucosidase Alfa 40 mg//kg | Cohort 3b: Alglucosidase Alfa in PAP | Total
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (3.4) | 8.1 (4.1) | 6.9 (2.7) | 4.7 (3.2) | 6.8 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 4 | 10
  Male | 5 | 3 | 2 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 3 | 2 | 3 | 4 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PAP: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious Treatment-emergent Adverse Events, and Adverse Event of Special Interest (AESI)
Description: Adverse event (AE): any untoward medical occurrence in participant received study drug & did not necessarily had to have causal relationship with treatment. TEAEs: AEs developed/worsened in grade/become serious during PAP period (from the time of 1st study drug dose up to Week 25). Serious AE(SAE): any untoward medical occurrence at any dose resulted in death, was life-threatening, required inpatient hospitalization, prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was medically important event. TEAEs included SAEs & non-SAEs. AESI:AE (serious/non-serious) of scientific & medical concern specific to Sponsor's product/program, for which ongoing monitoring & immediate notification by Investigator to Sponsor required.
Time Frame: From Baseline to Week 25
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg: Avalglucosidase alfa 20 mg/kg IV infusion qow for 25 weeks in PAP.
- PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg: Avalglucosidase alfa 40 mg/kg IV infusion qow for 25 weeks in PAP.
- PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg: After determination of the highest tolerated avalglucosidase alfa dose in Cohort 1 and Cohort 2 (after at least 5 participants in each Cohort 1 and Cohort 2 had received the 7th dose of avalglucosidase alfa or completed Week 13 with a minimum of 6 infusions), participants received avalglucosidase alfa 40 mg/kg (the highest tolerated dose) IV infusion qow for 25 weeks in PAP.
- PAP: Cohort 3b: Alglucosidase Alfa: After determination of the highest tolerated avalglucosidase alfa dose in Cohort 1 and Cohort 2 (after at least 5 participants in each Cohort 1 and Cohort 2 had received the 7th dose of avalglucosidase alfa or completed Week 13 with a minimum of 6 infusions), participants received alglucosidase alfa at their current stable dose (defined as dose [between 20 mg/kg qow and 40 mg/kg weekly as per physician] administered regularly for a minimum of 6 months immediately prior to entry in this study) IV infusion for 25 weeks in PAP.
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
Participants
  Any TEAEs | 5 | 5 | 5 | 5
  Any Serious TEAEs | 1 | 3 | 0 | 2
  Any AESI | 0 | 2 | 1 | 1

2. Primary Outcome: PAP: Number of Participants With Infusion-associated Reactions (IARs)
Description: IARs were defined as AESIs that occurred during either the infusion or the observation period following the infusion which were deemed to be related or possibly related to the study drug. Protocol-defined IARs: An AESIs that occurred during either the infusion or the observation period following the infusion which were deemed to be related or possibly related to study drug. Algorithm-defined IARs: any TEAE meeting either 1 or 2 criteria: 1) event occurred from the start of infusion to the end of infusion plus 24 hours, and considered related to study drug, 2) If an AE time component was missing, compared AE Start date with infusion start date and infusion end date. If an AE Start date was between infusion start date and infusion end date plus one day, and it was related to study drug.
Time Frame: From Baseline to Week 25
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
Participants
  Protocol-defined IARs | 0 | 2 | 1 | 1
  Algorithm-defined IARs | 0 | 2 | 1 | 1

3. Secondary Outcome: PAP: Number of Participants With Anti-drug Antibody (ADA) Response
Description: Anti-drug antibody response was categorized as: Treatment induced ADAs: ADAs developed de novo (seroconversion) following administration of study drug. Treatment boosted ADAs: pre-existing ADAs that were boosted at least two titer steps from Baseline (i.e., 4-fold increase in titers) followed by administration of study drug.
Time Frame: From Baseline to Week 25
Population: Analysis was performed on the ADA evaluable population which included participants who had received at least 1 infusion (partial or total) and had at least one ADA sample taken post-baseline after drug administration that was appropriate for ADA testing with a reportable result.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
Participants
  Treatment boosted ADA response | 0 | 0 | 1 | 2
  Treatment induced ADA response | 0 | 1 | 3 | 1

4. Secondary Outcome: PAP: Pharmacokinetic (PK) Parameter: Maximum Observed Plasma Concentration (Cmax) of Avalglucosidase Alfa
Description: Cmax is the maximum observed plasma concentration.
Time Frame: Cohort 1: pre-dose; at end of infusion; and at 2, 4, 6, and 8 hours after end of infusion on Day 1 (Week 1) and Week 25 Cohort 2 and 3: pre-dose; at end of infusion; and at 2, 4, 6, 8, and 12 to 16 hours after end of infusion on Day 1 (Week 1) and Week 25
Population: Analysis was performed on PK population which included PAP participants who had received at least 1 infusion (partial or total) and had evaluable drug concentration data. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for PAP: Cohort 3b: Alglucosidase Alfa arm.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
nanograms per milliliter
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 189000 (56700) | 403000 (171000) | 250000 (45100)
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 175000 (65900) | 297000 (60100) | 356000 (84700)

5. Secondary Outcome: PAP: Pharmacokinetic Parameter: Time to Achieve Maximum Observed Plasma Concentration (Tmax) of Avalglucosidase Alfa
Description: Tmax is the time to achieve maximum plasma concentration.
Time Frame: as for outcome 4
Population: Analysis was performed on PK population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for PAP: Cohort 3b: Alglucosidase Alfa arm.
Measure: Median (Full Range); unit: hours
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
hours
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 4.43 [3.90 to 5.33] | 7.00 [6.00 to 7.25] | 6.83 [6.65 to 7.22]
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 3.97 [3.77 to 4.75] | 7.13 [5.67 to 7.98] | 6.87 [5.03 to 7.43]

6. Secondary Outcome: PAP: Pharmacokinetic Parameter: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-last) of Avalglucosidase Alfa
Description: AUC0-last is the area under the plasma concentration versus time curve from time 0 to the time of last quantifiable concentration.
Time Frame: Cohort 1: pre-dose; at end of infusion; and at 2, 4, 6, and 8 hours after end of infusion on Day 1 (Week 1) and Week 25 Cohort 2 & 3: pre-dose; at end of infusion; and at 2, 4, 6, 8, and 12 to 16 hours after end of infusion on Day 1 (Week 1) and Week 25
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanograms*hours per milliliter
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
nanograms*hours per milliliter
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 923000 (352000) | 2630000 (972000) | 1720000 (255000)
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 805000 (295000) | 1930000 (348000) | 2200000 (533000)

7. Secondary Outcome: PAP: Pharmacokinetic Parameter: Terminal Half-life (t1/2) of Avalglucosidase Alfa
Description: t1/2 is the time required for the plasma concentration of a drug to decrease by half of its initial concentration.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
hours
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 0.703 (0.291) | 1.15 (0.523) | 0.806 (0.248)
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 0.601 (0.256) | 1.04 (0.248) | 1.19 (0.472)

8. Secondary Outcome: PAP: Pharmacokinetic Parameter: Clearance (CL) of Avalglucosidase Alfa
Description: CL is defined as a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters per hours
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
milliliters per hours
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 673 (222) | 562 (152) | 529 (150)
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 696 (203) | 683 (345) | 526 (125)

9. Secondary Outcome: PAP: Pharmacokinetic Parameter: Volume of Distribution at Steady State (Vss) of Avalglucosidase Alfa
Description: Steady state volume of distribution (Vss) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg
Number analyzed (Participants) | 6 | 5 | 5
milliliters
  Week 1: number analyzed (Participants) | 5 | 4 | 4
  Week 1 | 3550 (927) | 4500 (882) | 4300 (1420)
  Week 25: number analyzed (Participants) | 5 | 5 | 5
  Week 25 | 3520 (1180) | 5350 (2270) | 4020 (1390)

10. Secondary Outcome: PAP: Change From Baseline in Gross Motor Function Measure-88 (GMFM-88) Test Scores at Week 25
Description: GMFM-88 was developed specifically to detect quantitative changes in gross motor function. The GMFM-88 consisted of 88 items organized into 5 dimensions; lying and rolling (17 items); sitting (20 items); crawling and kneeling (14 items); standing (13 items) and walking, running and jumping (24 items). Each item was scored on a 4-point Likert scale with scores range: 0= cannot do; 1 = initiates less then [<] 10 percentage [%] of the task; 2 = partially completes [10% to <100% of the task] and 3 = task completion. The score for each dimension was expressed as a % of the maximum score for that dimension.Total percentage score was obtained by adding the percentage scores for each dimension and dividing the sum by the total number of dimensions. Total scores ranged from 0% to 100%; where higher scores indicated better motor functions.
Time Frame: Baseline, Week 25
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data for this OM.
Measure: Mean (Standard Deviation); unit: percentage of total score
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 4 | 6
percentage of total score | 6.50 (22.24) | 9.80 (13.99) | 11.00 (10.80) | 17.00 (8.44)

11. Secondary Outcome: PAP: Number of Participants in Gross Motor Function Classification System-Expanded and Revised (GMFCS-E and R) Scores at Baseline and Week 25
Description: GMFCS-E&R was a 5 level classification system for specific age ranges; observations were performed on 5 levels based on self-initiated movement, with emphasis on sitting, transfers, and mobility: Level I (walks without limitations), Level II (walks with limitations), Level III (walks using a hand-held mobility device), Level IV (self-mobility with limitations; may use powered mobility) and level V (transported in a manual wheel chair) (I to V). The distinctions between levels were based on functional limitations, the need for assistive mobility devices, and to a much lesser extent, quality of movement, and were designed to be meaningful in daily life. The lower level represented good motor functioning and higher level represented low motor functioning. Number of participants in each level of classification at Baseline and Week 25 were reported.
Time Frame: Baseline, Week 25
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
Participants
  Baseline: Level I | 1 | 1 | 2 | 3
  Baseline: Level II | 1 | 2 | 1 | 0
  Baseline: Level III | 1 | 0 | 1 | 1
  Baseline: Level IV | 2 | 2 | 0 | 1
  Baseline: Level V | 1 | 0 | 1 | 1
  Week 25: Level I | 1 | 1 | 2 | 3
  Week 25: Level II | 1 | 2 | 1 | 0
  Week 25: Level III | 2 | 1 | 0 | 1
  Week 25: Level IV | 1 | 1 | 1 | 1
  Week 25: Level V | 1 | 0 | 1 | 1

12. Secondary Outcome: PAP: Change From Baseline in Pompe Pediatric Evaluation of Disability Inventory (Pompe-PEDI) Functional Skills Scale: Mobility Domain Test Score-Scaled Score at Week 25
Description: Pompe-PEDI: disease specific version to assess functional capabilities and performance in children with Pompe disease from 2 months through adolescence. It comprised of Functional Skills Scale and Caregiver Assistance Scale; both scales had 3 domains: Self Care, Mobility, and Social Function. Mobility domain was used to measure change in mobility due to changes in muscle strength; consisted of 160 mobility items for participant/legal guardian. The total number of mobility items the child was capable of, was converted to a scaled score with a range of 0 to 100, where scores near "0" indicated low capability and scores near "100" indicated high capability), where higher score was indicative of greater functional ability. Scaled scores were used to interpret individual function and progress over time.
Time Frame: Baseline, Week 25
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 3 | 6
score on a scale | 6.19 (10.55) | 2.12 (4.04) | 2.60 (1.72) | 5.20 (5.95)

13. Secondary Outcome: PAP: Change From Baseline in Quick Motor Function Test (QMFT) Scores at Week 25
Description: QMFT was observer administered test comprised of 16 items specifically difficult for participants with Pompe disease. Each item was scored on 5-point ordinal scale ranged from 0 to 4 (higher score indicated better outcome). Total QMFT score was obtained by adding the scores of all items and ranged from 0 (unable to perform motor function tests) to 64 (normal muscle function), where higher score indicated better outcome/greater motor function.
Time Frame: Baseline, Week 25
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 4 | 6
score on a scale | -0.17 (4.45) | 3.20 (4.55) | 4.25 (3.30) | 5.17 (4.54)

14. Secondary Outcome: PAP: Echo-Left Ventricular Mass Z-Score (LVM Z-score) M-mode at Baseline, Week 25, and Change From Baseline at Week 25
Description: Cardiac function was evaluated using LVM Z-score as assessed by echocardiogram in M-mode. Z-Scores indicated the number of standard deviations (SD) from the mean in a normal distribution. The normal range is -2 to 2 and greater than 2 may indicate left ventricular hypertrophy. A negative change from Baseline indicated a decrease and positive change from Baseline indicated an increase in LVM Z-score. In this OM, absolute scores at Baseline and Week 25 along with Change from Baseline at Week 25 in LVM Z-score were reported.
Time Frame: Baseline, Week 25
Population: Analysis was performed on safety population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
Z-score
  Baseline: number analyzed (Participants) | 6 | 3 | 5 | 4
  Baseline | -1.10 (1.07) | 0.13 (2.39) | -0.78 (0.70) | -0.43 (0.92)
  Week 25: number analyzed (Participants) | 5 | 4 | 5 | 4
  Week 25 | -1.74 (2.01) | -1.05 (2.61) | -1.36 (0.99) | 0.15 (1.07)
  Change from Baseline at Week 25: number analyzed (Participants) | 5 | 2 | 5 | 3
  Change from Baseline at Week 25 | -0.60 (2.16) | -0.60 (0.71) | -0.58 (0.76) | 0.47 (1.76)

15. Secondary Outcome: PAP: Change From Baseline in Eyelid Position Measurements: Interpalpebral Fissure Distance (IPFD) - Left Non-Flash and Right Non-Flash at Week 25
Description: IPFD is the widest vertical distance (in millimeters) between the upper eyelid and the lower eyelid when the participant is looking in "primary gaze" (i.e. normal gaze when looking straight forward). Images were taken while the participants was wearing a pair of empty eyeglass frames with millimeters rulers attached as a standardized tool to measure eyelid position without camera flash. A negative change from Baseline indicated a decrease and positive change from Baseline indicated an increase in measured distance.
Time Frame: Baseline, Week 25
Population: Analysis was performed on safety population.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
millimeters
  Left non-Flash | -0.67 (1.54) | 1.30 (1.48) | 1.30 (0.76) | -0.50 (0.77)
  Right non-Flash | -0.92 (1.66) | 0.70 (1.25) | 0.90 (1.14) | -0.25 (1.13)

16. Secondary Outcome: PAP: Change From Baseline in Eyelid Position Measurements: Left and Right Margin Reflex Distance (MRD) at Week 25
Description: The MRD is the vertical distance (in millimeters) between the light reflex and the upper eyelid when the participant was looking in "primary gaze" while fixating on a light source. Images were taken while the participants was wearing a pair of empty eyeglass frames with millimeters rulers attached as a standardized tool to measure eyelid position. A negative change from Baseline indicated a decrease and positive change from Baseline indicated an increase in measured distance.
Time Frame: Baseline, Week 25
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
millimeters
  Left MRD: number analyzed (Participants) | 6 | 4 | 4 | 6
  Left MRD | -0.08 (1.53) | -0.38 (0.85) | 0.88 (1.11) | 0.08 (0.74)
  Right MRD: number analyzed (Participants) | 6 | 5 | 4 | 6
  Right MRD | -0.50 (1.61) | -0.50 (1.27) | 0.63 (1.03) | -0.08 (0.74)

17. Secondary Outcome: PAP: Change From Baseline in Eyelid Position Measurements Assessed by Margin Pupil Distance (MPD) - Left Non-Flash and Right Non-Flash at Week 25
Description: The MPD is the vertical distance (in millimeters) between the center of the pupil and the upper eyelid margin. Images were taken while the participants was wearing a pair of empty eyeglass frames with millimeters rulers attached as a standardized tool to measure eyelid position without camera flash. A negative change from Baseline indicated a decrease and positive change from Baseline indicated an increase in measured distance.
Time Frame: Baseline, Week 25
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
millimeters
  MPD Left Non-Flash: number analyzed (Participants) | 6 | 4 | 5 | 6
  MPD Left Non-Flash | -0.83 (1.44) | 0.75 (1.19) | 0.40 (0.42) | -0.50 (0.32)
  MPD Right Non-Flash | -0.25 (1.41) | 0.50 (1.06) | 0.30 (0.91) | 0.00 (0.71)

18. Secondary Outcome: PAP: Change From Baseline in Creatine Kinase Value at Week 25
Description: Change from Baseline in Creatine kinase value (to assess muscle damage) at Week 25 were reported in this OM.
Time Frame: Baseline, Week 25
Population: Analysis was performed on safety population.
Measure: Mean (Standard Deviation); unit: international units per liters
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa
Number analyzed (Participants) | 6 | 5 | 5 | 6
international units per liters | -208.67 (382.34) | -476.60 (467.20) | -421.40 (413.39) | -1.33 (51.20)

19. Secondary Outcome: ETP: Number of Participants With Treatment Emergent Adverse Events, Serious Treatment Emergent Adverse Events, and Adverse Event of Special Interest
Description: Data for this outcome measure will be reported at the time of anticipated last participant last visit results posting (August 2028).
Time Frame: Up to 9 years and 4 months
Reporting Status: Not Posted, anticipated posting 2028-08

20. Secondary Outcome: ETP: Number of Participants With Infusion-associated Reactions
Description: as for outcome 19
Time Frame: Up to 9 years and 4 months
Reporting Status: Not Posted, anticipated posting 2028-08

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 25 in PAP and from Week 26 to 102 in ETP. Safety data were planned to be collected and analyzed for pooled population of participants who received avalglucosidase alfa 40 mg/kg (Cohorts 2 and 3a of PAP) in ETP. AE data collection is still ongoing and will be updated upon study completion.
Description: TEAEs: AEs that developed/worsened in grade/become serious during treatment epoch (for PAP:time just prior to 1st study drug dose in ETP or 4 weeks after last infusion for those who didn't get into ETP or 2 weeks after last infusion in PAP if participant enrolled in another study/received ERT) (for ETP:time from 1st administration of study drug in ETP to last administration of study drug +4 weeks /2 weeks if participant got enrolled in another study/received ERT). Analyzed on safety population.
Groups:
- ETP: Avalglucosidase Alfa 20 mg/kg: Included all participants of Cohort 1 who received avalglucosidase alfa 20 mg/kg IV infusion qow for 25 weeks in PAP, followed by same treatment from Week 26 up to Week 371 in ETP.
- Pooled Arm ETP: Avalglucosidase Alfa 40 mg/kg: Pooled arm included all participants of Cohorts 2 and 3a who received avalglucosidase alfa 40 mg/kg IV infusion qow for 25 weeks in PAP, followed by same treatment from Week 26 up to Week 371 in ETP.
- Alglucosidase Alfa in PAP Then Avalglucosidase Alfa 40 mg/kg in ETP: Included all participants of Cohort 3b who received alglucosidase alfa at their current stable dose (defined as dose [between 20 mg/kg qow and 40 mg/kg weekly as per physician] administered regularly for a minimum of 6 months immediately prior to entry in this study) IV infusion for 25 weeks in the PAP and after PAP, switched to receive avalglucosidase alfa 40 mg/kg IV infusion qow from Week 26 up to Week 371 in ETP.
Arm/Group | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg | PAP: Cohort 3b: Alglucosidase Alfa | ETP: Avalglucosidase Alfa 20 mg/kg | Pooled Arm ETP: Avalglucosidase Alfa 40 mg/kg | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa 40 mg/kg in ETP
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/6 | 0/6 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/5 | 0/5 | 2/6 | 4/6 | 2/10 | 1/3
Other Adverse Events (participants affected / at risk) | 5/6 | 5/5 | 5/5 | 4/6 | 6/6 | 7/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg (N=6) | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg (N=5) | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg (N=5) | PAP: Cohort 3b: Alglucosidase Alfa (N=6) | ETP: Avalglucosidase Alfa 20 mg/kg (N=6) | Pooled Arm ETP: Avalglucosidase Alfa 40 mg/kg (N=10) | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa 40 mg/kg in ETP (N=3)
Atrial Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid Ptosis (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Infection Pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device Malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Cohort 1: Avalglucosidase Alfa 20 mg/kg (N=6) | PAP: Cohort 2: Avalglucosidase Alfa 40 mg/kg (N=5) | PAP: Cohort 3a: Avalglucosidase Alfa 40 mg/kg (N=5) | PAP: Cohort 3b: Alglucosidase Alfa (N=6) | ETP: Avalglucosidase Alfa 20 mg/kg (N=6) | Pooled Arm ETP: Avalglucosidase Alfa 40 mg/kg (N=10) | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa 40 mg/kg in ETP (N=3)
Lymph Node Pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerumen Impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive Cerumen Production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Middle Ear Effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivochalasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental Caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (4) | 1 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces Soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loose Tooth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucous Stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (6) | 0 (0) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 2 (2) | 3 (3) | 1 (3) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter Site Oedema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device Related Thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Site Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 1 (4) | 2 (2) | 1 (1) | 2 (9) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Bronchitis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Infection Pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis Externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stoma Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (5) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Viral Rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha-1 Acid Glycoprotein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecal Calprotectin Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (14) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enuresis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staring (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurogenic Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital Erosion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 1 (13) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Pulmonary Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia Areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 1 (1) | 2 (3) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03019406/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03019406/SAP_001.pdf